CLINICAL TRIAL: NCT05341557
Title: A Phase 1 Open-label Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of BPI-371153 in Subjects with Advanced Solid Tumors or Relapsed/Refractory Lymphoma
Brief Title: A Phase 1 Study of BPI-371153 in Subjects with Advanced Solid Tumors or Relapsed/Refractory Lymphoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Betta Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BTP-661611
Record Dates: First submitted 2022-04-18; First posted 2022-04-22 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Advanced Solid Tumor; Lymphoma; NSCLC; HCC
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dose Escalation (Experimental): Oral capsules taken in escalating levels to determine MTD/RP2D. Each treatment cycle will be 21 days in duration with BPI-371153 administered, once daily (QD).
  Interventions: Drug: BPI-371153
- Dose Expansion (Experimental): Oral capsules administered at recommended doses. Each treatment cycle will be 21 days in duration with BPI-371153 administered, once daily (QD).
  Cohort 1: Advanced NSCLC Cohort 2: Relapsed/refractory lymphoma Cohort 3: Advanced HCC Cohort 4: Other Advanced Solid Tumors
  Interventions: Drug: BPI-371153

INTERVENTIONS:
Drug: BPI-371153 — Subjects will receive BPI-371153 until disease progression

SUMMARY:
A first-in-human study to evaluate the safety, tolerability and maximum tolerated dose (MTD) and establish the recommended phase 2 dose (RP2D) of BPI-371153, a PD-L1 Inhibitor, in patients with advanced solid tumors or relapsed/refractory lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Dose escalation phase: Age ≥18 and ≤65 years, male and female patients; Dose expansion phase: Age ≥18, male and female patients;
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-1;
* Dose escalation phase: histologically or cytologically confirmed locally advanced or metastatic solid tumor patients (excluding HCC patients) or relapsed/refractory lymphoma, who had disease progression after standard therapy, intolerable to standard therapy, refuse to standard therapy or for whom no standard therapy exists;
* Dose expansion phase: histologically or cytologically confirmed locally advanced or relapsed/metastatic Non-Driver Mutation NSCLC, relapsed/refractory lymphoma, HCC with Child-Pugh A or B(≤ 7 points), or other diagnosed solid tumor patients who had disease progression after standard therapy, intolerable to standard therapy, refuse to standard therapy or for whom no standard therapy exists;
* Evaluable lesion required for dose escalation phase and at least 1 measurable lesion as per RECIST v1.1( for other diagnosed solid tumos excluding HCC), mRECIST(for HCC) or Lugano 2014(for lymphoma);
* Adequate organ function;

Exclusion Criteria:

* Dose escalation phase: Prior immune checkpoint inhibition with anti-programmed cell death-1 (PD1)/programmed death ligand-1(PD-L1) or programmed death ligand-2(PD-L2) therapy;
* Dose expansion phase: Prior immune checkpoint inhibition with anti-programmed cell death-1 (PD1)/programmed death ligand-1(PD-L1) or programmed death ligand-2(PD-L2) therapy within 28 days prior to treatment. Subjects with a history of a Grade 3 or higher immune-related AE from prior immunotherapies;
* Prior other specific T cell targeting agents;
* Use of systemic or absorbable topical corticosteroids therapy(≥ 10 mg/day prednisone or equivalent) two weeks prior to start of treatment.
* Inadequate wash-out of prior therapies described per protocol, which may include anti-tumor therapies, tumor adjuvant drugs, organ or stem cell transplantation, moderate or strong CYP3A inhibitor or inducer, and vaccine;
* Patients with major surgery within 4 weeks, severe or unstable systemic disease, unstable/symptomatic CNS metastasis, other malignant tumors, autoimmune disease, ILD, clinical significant cardiac disease, bleeding or embolic disease, active infectious disease, conditions affecting drug swallow and absorption, medical history leading to chronic diarrhea, etc;
* Pregnancy or lactation;
* Other conditions considered not appropriate to participate in this trial by the investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2022-08-29 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
The adverse events (AEs) | Through the Phase I, approximately 24 months
  Safety and tolerability will be assessed by monitoring frequency, duration and severity of adverse events (AEs)
Determine the recommended Phase II dose (RP2D) | Through the Phase I, approximately 24 months
  Number of subjects with dose limiting toxicity

SECONDARY OUTCOMES:
Evaluate the pharmacokinetics of BPI-371153 | Through the Phase I, approximately 24 months
  Based on blood plasma concentration
Determination of anti-tumor activity of BPI-371153 | Through the Phase I, approximately 24 months
  Efficacy assessments (tumor evaluation) will be performed per RECIST1.1, mRECIST or Lugano 2014 depending on tumor type.
To explore the levels of expression of PD-L1 associated with BPI-371153 clinical activity | Through the Phase I, approximately 24 months
  Based on the levels of expression of PD-L1 and anti-tumor activity of BPI-371153

CONTACTS AND LOCATIONS:
Overall Officials: Yuankai Shi, Ph.D, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (4):
- China (4):
  - Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Chaoyang, Beijing Municipality
  - Cangzhou Central Hospital, Cangzhou, Hebei
  - Tianjin Cancer Hospital, Tianjin, Tianjin Municipality
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No